CLINICAL TRIAL: NCT03219372
Title: Pravastatin Intervention to Delay Hepatocellular Carcinoma Recurrence
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study discontinued due to low accrual.
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Shehnaz Hussain, Associate Professor, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IIT2017-08-HUSSAIN-STATLV; 1R01CA218486-01 (NIH)
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-12

CONDITIONS: Hepatocellular Carcinoma; Liver Cirrhoses
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Pravastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Intervention Model Description: 1:1 drug versus placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pravastatin Pill (Experimental): Daily pravastatin (40mg)
  Interventions: Drug: Pravastatin Pill
- Placebo Oral Tablet (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Pravastatin Pill — statin
  Other Names: statin
  Arms: Pravastatin Pill
Drug: Placebo Oral Tablet — placebo
  Other Names: placebo
  Arms: Placebo Oral Tablet

SUMMARY:
Hepatocellular Carcinoma (HCC) is a major health concern in the United States, particularly among people with liver cirrhosis. Out of every 100 patients with liver cancer, only 18 will survive 5 years or more. While locoregional therapies are utilized in an effort to combat this disease, the recurrence rate of HCC after these therapies are high.

Statins are widely used drugs that lower cholesterol levels. Some studies have suggested that statins lower risk of HCC recurrence, but this possibility has not been studied thoroughly in a clinical trial. This study will examine the effects of pravastatin, a type of statin, on time to HCC recurrence in patients with early stage HCC. It is possible that pravastatin in combination with locoregional therapies may delay or protect against HCC recurrence.

DETAILED DESCRIPTION:
To date, there has been a scarcity of clinical trials evaluating the effectiveness of adjuvant therapies in patients with early stage HCC, although it is widely considered an area of highly unmet need.

The objective of this randomized double-blinded, placebo-controlled Phase II trial is to examine the effects of pravastatin use versus placebo after 12 months of treatment on hepatocellular cancer (HCC) recurrence in 130 patients with liver cirrhosis, HCC meeting Milan Criteria or OPTN tumor downstaging criteria for tumor burden, and initial locoregional therapy (LRT) with adequate response.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Confirmed diagnosis of liver cirrhosis (Child-Pugh A or B) assessed by the presence of clinical signs, symptoms, body imaging, or liver biopsy
* Diagnosis of HCC falling within one of the following criteria prior to LRT. Criteria fulfillment will be confirmed by the Imaging Charter and MedQIA.

  1. One lesion ≤ 5 cm or two to three lesions, each ≤ 3 cm.
  2. One lesion > 5 cm and ≤ 8 cm.
  3. Two or three lesions, of which at least one is > 3 cm and all are ≤ 5 cm each. The sum of all diameters must be ≤ 8 cm.
  4. Four or five lesions, each < 3 cm. The sum of all diameters must be ≤ 8 cm.
* Initiation of LRT (according to clinical judgement) within 24 months prior to Screening Visit, with adequate response as determined by Imaging Charter and MedQIA.
* ECOG performance status ≤1 (Karnofsky ≥70%; see Appendix A)
* AST (SGOT) & ALT (SGPT) ≤5 × institutional ULN
* AFP < 400 ng/mL
* Ability to understand and the willingness to sign a written informed consent document and medical release
* Agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; for women who are able to become pregnant.
* Willing and able to comply with trial protocol and follow-up

Exclusion Criteria:

* Current use of statin medication or statin use within 12 months of Screening visit.
* Current systemic use of medications known to interact with statins and potentially increase toxicity, including (e.g., gemfibrozil, cyclosporine, clarithromycin, colchicine, niacin and fibrates).
* History of adverse effects, intolerance, or allergic reactions attributed to compounds of similar chemical or biologic composition to pravastatin (i.e., other statin medications)
* Current use of any other investigational agents
* Women who are pregnant. Women who are able to become pregnant must have a confirmed negative pregnancy test prior to enrollment.
* Women who are breastfeeding. It is not known whether pravastatin is excreted into human milk; however, a small amount of another drug in this class does pass into breast milk. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pravastatin, breastfeeding should be discontinued if the mother is treated with pravastatin.
* Prior liver transplant
* MELD score ≥30.
* History of chronic myopathy
* Active malignancy within the past 5 years (excluding HCC, basal/squamous cell skin cancer, or prostate cancer with a Gleason score 6 or less)
* Known HIV infection
* Hemophilia
* Concurrent illness which in the opinion of the investigators would compromise either the patient or the integrity of the data
* Concurrent excessive alcohol consumption (average alcohol consumption of more than 5 drinks per day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2019-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shehnaz Hussain, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pravastatin Pill: Pravastatin 40 mg, daily for 12 months
  Pravastatin, a lipid-lowering agent, is a derivative of ML236B (compactin), which was identified in a fungus called Penicillium citrinum in the 1970s. It is an inhibitor of 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase.
- Placebo Oral Tablet: Placebo identical in color, consistency, and appearance to pravastatin 40 mg, daily for 12 months
  Placebo: A substance that has no therapeutic effect, and will be used as a control in testing the study agent.
Period: Overall Study
Arm/Group | Pravastatin Pill | Placebo Oral Tablet
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: 0 participants enrolled in placebo group due to 1 total participant enrollment in pravastatin group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pravastatin Pill | Placebo Oral Tablet | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 1 |  | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 1 |  | 1
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 0 |  | 0
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Recurrence
Description: Mean difference in time (in months) from baseline (study visit 1) to first hepatocellular cancer (HCC) recurrence or HCC death within 12 months following treatment initiation for subjects randomized to pravastatin versus subjects randomized to placebo.
  - HCC recurrence will be confirmed by central expert independent radiographic review.
Time Frame: 12 months from baseline
Population: As accrual fell far below target, for associated privacy considerations related to the potential for participant re-identification, data are not reported.
Arm/Group | Pravastatin Pill | Placebo Oral Tablet
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Recurrence Free Survival
Description: Mean difference in time (in months) from baseline (study visit 1) to first occurrence of a documented hepatocellular cancer (HCC) recurrence within 12 months following treatment initiation for subjects randomized to pravastatin versus subjects randomized to placebo.
  - HCC recurrence will be confirmed by central expert independent radiographic review.
Time Frame: 12 months from baseline
Population: as for outcome 1
Arm/Group | Pravastatin Pill | Placebo Oral Tablet
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Survival
Description: Mean difference in time (in months) from baseline (study visit 1) to death (for any reason) within 12 months following treatment initiation for subjects randomized to pravastatin versus subjects randomized to placebo.
Time Frame: 12 months from baseline
Population: as for outcome 1
Arm/Group | Pravastatin Pill | Placebo Oral Tablet
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Waitlist Drop-off
Description: Mean difference in time from baseline (study visit 1) to liver transplant waitlist drop-off within 12 months following treatment initiation for subjects randomized to pravastatin versus subjects randomized to placebo.
Time Frame: 12 months from baseline
Population: as for outcome 1
Arm/Group | Pravastatin Pill | Placebo Oral Tablet
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Liver Stiffness
Description: Mean difference in mean change in liver stiffness (as measured by MRE or FibroScan) between baseline (study visit 1) and 12 months (study visit 6) for subjects randomized to pravastatin versus subjects randomized to placebo.
Time Frame: 12 months from baseline
Population: as for outcome 1
Arm/Group | Pravastatin Pill | Placebo Oral Tablet
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Liver Fat Fraction
Description: Mean difference in within-person change in liver fat fraction (as measured by MRE) between baseline (study visit 1) and 12 months (study visit 6) for subjects randomized to pravastatin versus subjects randomized to placebo.
Time Frame: 12 months from baseline
Population: as for outcome 1
Arm/Group | Pravastatin Pill | Placebo Oral Tablet
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Serum Biomarkers of Monocyte/Macrophage and Stellate Cell Activation
Description: Mean difference in serum biomarkers including cytokines, chemokines, soluble receptors, and proteins (eg. IL6, TNFα, sTNFRII, IL18BP, sCD163, IL10, IL17, IL-8, CCL17, TGFβ) from baseline (study visit 1) to 12 months (study visit 6) for subjects randomized to pravastatin versus subjects randomized to placebo.
Time Frame: 12 months from baseline
Population: as for outcome 1
Arm/Group | Pravastatin Pill | Placebo Oral Tablet
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Levels of Liver Tissue Markers Related to HCC
Description: Mean difference in liver tissue markers related to HCC including those in the Wnt/β-catenin pathway (eg. β-catenin, glutamine synthetase) from baseline (study visit 1) to 12 months (study visit 6) for subjects randomized to pravastatin versus subjects randomized to placebo.
Time Frame: 12 months from baseline
Population: as for outcome 1
Arm/Group | Pravastatin Pill | Placebo Oral Tablet
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 2-month* intervention period (one patient and early withdrawal at Visit 2) and within 90 days after the last administration of the study drug. *Scheduled intervention period for this study was 12 months with 6 study visits.
Description: Regular investigator assessment, regular laboratory testing, self-reporting.
Arm/Group | Pravastatin Pill | Placebo Oral Tablet
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pravastatin Pill (N=1) | Placebo Oral Tablet (N=0)
Fatigue (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Accrual fell well below target. One subject was randomized to the study and withdrew prior to completion. Outcome measures were not analyzed due to insufficient accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/72/NCT03219372/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/72/NCT03219372/ICF_001.pdf